CLINICAL TRIAL: NCT05921604
Title: Baclofen Versus Gabapentin in Preventing Postoperative Pain After Laparoscopic Sleeve
Brief Title: Baclofen Versus Gabapentin in Preventing Postoperative Pain After Laparoscopic Sleeve Gastrectomy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Gamal Moussa, Assistant Lecturer at Clinical Pharmacy department , Faculty of Pharmacy -Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 35648
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-11

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Baclofen; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (baclofen) (Experimental): which will include 50 patients scheduled for sleeve gastrectomy and will receive 10 mg oral baclofen 1 h before anesthesia.
  Interventions: Drug: Baclofen 10mg
- Group 2 (gabapentin) (Experimental): which include 50 patients scheduled for sleeve gastrectomy and will receive 600 mg oral gabapentin 1 h before anesthesia.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Baclofen 10mg — which will include 50 patients scheduled for sleeve gastrectomy and will receive 10 mg oral baclofen 1 h before anesthesia.
  Arms: Group 1 (baclofen)
Drug: Gabapentin — which include 50 patients scheduled for sleeve gastrectomy and will receive 600 mg oral gabapentin 1 h before anesthesia.
  Arms: Group 2 (gabapentin)

SUMMARY:
The aim of this study is to compare the possible efficacy of baclofen and gabapentin on postoperative pain in patient with morbid obesity who will undergo laparoscopic sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* - Age between 18-60 years old.
* Both male and female patients will be included.
* Morbidly obese patients scheduled for sleeve gastrectomy with BMI ≥35 kg/m2 with the presence of comorbidity such as hypertension, arthritis, and diabetes.
* Morbidly obese patients scheduled for sleeve gastrectomy with BMI ≥ 40 kg/m2 without comorbidity.
* Patients fit for anesthesia and surgery.

Exclusion Criteria:

* Patients with BMI >55 kg/m2.
* Patients with previous procedures for the treatment of obesity.
* Pregnant females and lactating women.
* Patients with psychological or psychiatric disease
* Administration of antiemetic medication or systemic corticosteroids within 24 hours before surgery
* Patients who experienced vomiting within 24 hours before surgery.
* Patients with history of alcohol or drug abuse.
* Patients with hypersensitivity or contraindications to any of the drugs used in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) score | The first 48 hours after surgery.
  During the first 48-h postoperative study period, patients were asked to rate their intensity of pain using visual analog scale (VAS) scores. the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post-surgical patients (knee replacement, hysterectomy, or laparoscopic myomectomy who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
sedation score | The first 48 hours after surgery.
  Postoperative sedation scores will be evaluated using the following scale: 0 = awake, 1 = mild sedation, 2 = sleepy but arousable, and 3 = very sleepy.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal and Laparoscopic Surgery Unit, General Surgery Department, Tanta University Hospital, Tanta, Egypt, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No